CLINICAL TRIAL: NCT00182182
Title: Congestive Heart Failure Assessment and Management in Primary Care: CHAMP
Brief Title: Evaluation of a Primary Care Based Heart Failure Management Program
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: HSF2004h00511
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2006-09

CONDITIONS: Heart Failure
Keywords: Heart Failure; Family physicians; academic detailing; process of care
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Behavioral: Primary care based disease management strategy

SUMMARY:
Evaluation of a primary care based (family physicians) HF management strategy in patients with heart failure in the community

DETAILED DESCRIPTION:
Cluster randomized clinical trial (family physician is cluster) evaluating a primary care based heart failure management strategy

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age more or equal to 65 years AND
2. Diagnosis of HF confirmed with the following criteria:

   1. Previous hospital admission for HF OR
   2. Definite HF confirmed with the Boston HF criteria OR
   3. Possible HF confirmed with the Boston HF criteria AND evidence of left ventricular systolic dysfunction (left ventricular ejection function <40%) on echocardiography, radionuclide angiography, or left ventricular angiogram documented in the patient's family physicians clinic chart.

Exclusion Criteria:

1. Patients with terminal illness (e.g. cancer) with a life expectancy of less than one year.
2. Patients in a long-term-care facility with nursing care.
3. Patients awaiting cardiac surgery for correctable causes of HF (e.g., severe valvular disease or extensive ischemia) during the study period.
4. Patients expected to be away from the country during the intervention period for a duration of >3 months.
5. Patients unable or refusing to sign consent.
6. Patients currently followed in the Hamilton Health Sciences HF clinic. These patients are excluded as they are currently enrolled in a HF disease management strategy.
7. Patients currently enrolled in another clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170
Dates: Start 2003-07; Study Completion 2006-10

PRIMARY OUTCOMES:
Process-of-care composite score assessed at baseline, at 6 months for effectiveness of the intervention, and at 12 months for sustainability of the effect. The score includes assessment of:
ACE-inhibitor use unless contraindicated,ACE-inhibitor dosage is at >50% of clinical trial target dose,Beta-blocker use unless contraindicated.
Each component of the score will be given one point.

SECONDARY OUTCOMES:
Disease specific quality of life (QOL)with Minnessota Living with Heart Failure.
NYHA functional class.
Other outcomes
All-cause hospitalization defined as > 24-hour hospital stay including the time spent in the emergency room.
Hospitalizations for HF: > 24-hour hospital stay including the time spent in the emergency room with clinical evidence of HF including at least one of the following: increased dyspnea on exertion, orthopnea, nocturnal dyspnea, elevated jugular venous
Emergency room visits for deterioration of HF requiring IV or additional PO diuretics: <24-hour stay in hospital/emergency room with clinical evidence of HF.
Referral to Hamilton Health Sciences HF clinic or other institution.
Quality adjusted survival
Overall costs

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Demers, MD, MSc, FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada